CLINICAL TRIAL: NCT06912087
Title: A Phase I Study of Zanzalintinib With Pembrolizumab and Cetuximab in Patients With Recurrent and/or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Dose Finding Study of Zanzalintinib With Pembrolizumab and Cetuximab in Head and Neck SCC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB24-1994
Record Dates: First submitted 2025-01-31; First posted 2025-04-04 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Neoplasms; Carcinoma, Squamous Cell; Neoplasm Recurrence, Local; Neoplasm Metastasis; Recurrent Squamous Cell Carcinoma; Metastatic Squamous Cell Carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell; Neoplasm Recurrence, Local; Neoplasm Metastasis | interventions — Cetuximab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation (Dose Level -1) (Experimental): Participants receive the combination of the following drugs in 42-day cycles:
  * Zanzalintinib at a dose of 20 mg daily on days 1-42 of each cycle
  * Cetuximab at a dose of 500 mg/m2 on days 1, 15, and 29 of each cycle
  * Pembrolizumab 400 mg on day 1 of each cycle
  Interventions: Drug: Zanzalintinib; Drug: Cetuximab; Drug: Pembrolizumab
- Dose Escalation (Dose Level 0) (Experimental): Participants receive the combination of the following drugs in 42-day cycles:
  * Zanzalintinib at a dose of 40 mg daily on days 1-42 of each cycle
  * Cetuximab at a dose of 500 mg/m2 on days 1, 15, and 29 of each cycle
  * Pembrolizumab 400 mg on day 1 of each cycle
  This will be the first dose escalation enrolled. Dose Levels 1 and/or -1 will be enrolled depending on side effects seen in participants enrolled to this cohort.
  Interventions: Drug: Zanzalintinib; Drug: Cetuximab; Drug: Pembrolizumab
- Dose Escalation (Dose Level 1) (Experimental): Participants receive the combination of the following drugs in 42-day cycles:
  * Zanzalintinib at a dose of 60 mg daily on days 1-42 of each cycle
  * Cetuximab at a dose of 500 mg/m2 on days 1, 15, and 29 of each cycle
  * Pembrolizumab 400 mg on day 1 of each cycle
  Interventions: Drug: Zanzalintinib; Drug: Cetuximab; Drug: Pembrolizumab
- Dose Expansion (Experimental): Participants receive the combination of the following drugs in 42-day cycles:
  * Zanzalintinib will be dosed daily (days 1-42) at the dose identified as recommended phase 2 dose during dose escalation.
  * Cetuximab at a dose of 500 mg/m2 on days 1, 15, and 29 of each cycle
  * Pembrolizumab 400 mg on day 1 of each cycle
  The expansion cohort will begin enrollment after the dose escalation cohorts have completed enrollment.
  Interventions: Drug: Zanzalintinib; Drug: Cetuximab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Zanzalintinib — Experimental receptor tyrosine kinases (RTKs)
  Other Names: XL 092; XL-092; XL092
Drug: Cetuximab — Food and Drug Administration (FDA) approved monoclonal antibody directed against the epidermal growth factor (EGFR).
  Other Names: Erbitux
Drug: Pembrolizumab — FDA approved monoclonal immunoglobulin (Ig) G4 antibody directed against human cell surface receptor PD-1 (programmed death-1 or programmed cell death-1)
  Other Names: Keytruda

SUMMARY:
This Phase I clinical trial evaluates the safety, tolerability, and optimal dosing of Zanzalintinib in combination with Pembrolizumab and Cetuximab in patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck (R/M HNSCC). The study aims to establish the maximally tolerated dose (MTD) and recommended Phase II dose (RP2D) while also exploring efficacy outcomes, including progression-free survival (PFS) and overall survival (OS).

DETAILED DESCRIPTION:
This Phase I, single-site clinical trial investigates the combination therapy of Zanzalintinib, an oral tyrosine kinase inhibitor, with Pembrolizumab, an anti-PD1 immune checkpoint inhibitor, and Cetuximab, an anti-EGFR monoclonal antibody, in patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck (R/M HNSCC). The primary objective is to determine the maximally tolerated dose (MTD) and the recommended Phase II dose (RP2D) of Zanzalintinib in combination with Pembrolizumab and Cetuximab.

Secondary objectives include evaluating safety, tolerability, objective response rate (ORR), progression-free survival (PFS), and overall survival (OS). Exploratory objectives will investigate the effects of the treatment on plasma circulating tumor DNA (ctDNA) levels, immune phenotype, genetic alterations, and histopathologic changes in tumor biopsies.

The trial uses a dose-escalation design, with a 42-day treatment cycle, to assess safety and dose-limiting toxicities. This combination targets the immune-suppressive tumor microenvironment, aiming to overcome resistance mechanisms and improve clinical outcomes for a population with limited therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed recurrent and/or metastatic squamous cell carcinoma of the head and neck (R/M HNSCC), which is considered incurable by local therapies.
* Primary tumor locations: oropharynx, oral cavity, hypopharynx, larynx, nasopharynx, and sinonasal. Unknown primary is also eligible.
* Age: Participants must be at least 18 years old.
* ECOG Performance Status: Must be 0-1.
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
* For oropharyngeal cancer: HPV (p16) testing is required. p16 Immunohistochemistry (IHC) is sufficient for Human Papillomavirus (HPV) testing.
* Programmed cell death ligand 1 (PD-L1) combined positive score (CPS) : For patients with previously untreated R/M disease, a combined positive score (CPS) of 1 or greater is required. There is no PD-L1 restriction for patients who have previously received anti-PD(L)1 therapy.
* Recovery to baseline or ≤ Grade 1 severity (CTCAE v5) from any adverse events (AEs), including immune-related AEs from prior treatments.
* Adequate organ and marrow function, including:
* Absolute neutrophil count (ANC) ≥ 1500/mm3.
* Platelets ≥ 100,000/mm3.
* Hemoglobin ≥ 9 g/dL.
* Normal liver and kidney function.
* Capable of understanding and complying with the protocol requirements and must have signed the informed consent document.
* Contraception: Sexually active fertile subjects must agree to use a highly effective method of contraception during the study and for 2 months after the last dose of cetuximab and 4 months after the last dose of pembrolizumab.

Exclusion Criteria:

* Prior treatment with Zanzalintinib or other vascular endothelial growth factor receptor (VEGFR)-targeted therapies, -Cetuximab, or other epidermal growth factor receptor (EGFR) inhibitors.
* More than two prior lines of systemic therapy in the recurrent/metastatic setting.
* Relapsed disease within 3 months of definitive therapy.
* Prior treatment with small molecule kinase inhibitors, chemotherapy, biologic, or other anticancer therapies within certain time frames (2-4 weeks before the first dose of study treatment).
* Brain metastases or cranial epidural disease unless stable after treatment for at least 4 weeks.
* Concomitant anticoagulation with oral anticoagulants or platelet inhibitors, unless on stable doses of acceptable anticoagulants.
* Active infection requiring systemic treatment or significant cardiovascular, gastrointestinal, or other serious health issues that may affect study participation.
* Known or suspected autoimmune disease, except for specific conditions like type I diabetes or controlled skin disorders.
* Pregnancy or breastfeeding: Women must not be pregnant or breastfeeding at screening.
* Other malignancies within the past 2 years (except for certain low-grade cancers like localized skin cancers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2027-06-05 (Estimated); Study Completion 2027-06-05 (Estimated)

PRIMARY OUTCOMES:
Maximally Tolerated Dose (MTD) of Zanzalintinib in Combination with Pembrolizumab and Cetuximab | end of DLT evaluation period (first 28 days of treatment)
  The MTD will be defined as the dose combination with a dose-limiting toxicities (DLT) rate closest to the target DLT rate of 25%.
Recommended Phase II Dose (RP2D) of Zanzalintinib in Combination with Pembrolizumab and Cetuximab | End of enrollment
  The RP2D will be defined as the MTD identified after enrollment to all cohorts.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years from the date of the final subject accrual on study
  The secondary outcome measure of Progression-Free Survival (PFS) will assess the time from the first dose of the study drug (Zanzalintinib, Pembrolizumab, and Cetuximab) to the date of documented disease progression (PD) based on RECIST v1.1 or death, whichever occurs first. This measure will help evaluate the efficacy of the combination therapy in delaying disease progression in patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck.
Overall Survival (OS) | 2 years from the date of the final subject accrual on study
  The secondary outcome measure of Overall Survival (OS) will evaluate the time from the first dose of the study drug (Zanzalintinib, Pembrolizumab, and Cetuximab) to the date of death from any cause. This outcome will help assess the overall impact of the combination therapy on patient survival in recurrent and/or metastatic squamous cell carcinoma of the head and neck.
Safety of zanzalintinib in combination with pembrolizumab and cetuximab | End of treatment (about 24 months on average)
  Adverse events (AEs) leading to discontinuation or death, and severity of AEs will be assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ari Rosenberg, MD, Principal Investigator — University of Chicago Medicine Comprehensive Cancer Center
Locations (1):
- University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The document you provided does not include a specific IPD (Individual Patient Data) Sharing Plan or details regarding what patient data may be shared with other researchers. Typically, this information is outlined in separate documentation, such as consent forms or data sharing agreements, and would depend on institutional policies or specific regulatory requirements.
  If you require more detailed information about the plan to share IPD for this study, I recommend contacting the Principal Investigator or the University of Chicago Medicine Comprehensive Cancer Center directly to inquire about their data sharing practices.